CLINICAL TRIAL: NCT05556694
Title: Association Between Cumulative Fluids Balance and Ventilator Associated Events in Critically Ill Patients: a Prospective Cohort Study
Brief Title: Cumulative Fluids Balance and Ventilator Associated Events
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sahar Younes, Assistant professor, Damanhour University
Other Study IDs: ventilator associated events
Record Dates: First submitted 2022-09-17; First posted 2022-09-27 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Ventilator Associated Event
Keywords: Cumulative fluids balance; Ventilator Associated Event; Critically ill patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: calculation of cumulative fluid balance — - We will calculate cumulative fluid balance as daily fluid balance within four days of the event of interest. Cumulative fluid balance will be computed as the sum of daily fluid balances over the previous 24 hours, calculated by total fluid input minus total fluid output on a specific day of ICU admission over the first four calendar days of mechanical ventilation. Insensible fluid loss, such as perspiration or evaporative water loss related to respiration will not be routinely assessed and will not be included in the calculation of cumulative fluid balance. The cumulative fluid balance from day 0 to day 1 will be labelled as day 1, and the following days as day 2 and day 3. Cumulative fluid balance at day 3 refers to the cumulative fluid balance during the first four calendar days.
  Other Names: VAEs assessment

SUMMARY:
Fluid therapy is widely used to improve organ perfusion and survival in critically patients. Fluid therapy is an important component of intensive care management; however, optimal fluid management is unknown. Inadequate or excessive fluid resuscitation, on the other hand, is linked with a poor prognosis; the former can cause tissue hypo-perfusion and exacerbate organ dysfunction, while the latter can raise the risk of heart failure, pulmonary edema, and pleural effusions. Ventilator-associated lung injury (VALI) is a devastating complication of assisted mechanical ventilation (MV) and is one of the root causes of prolonged MV.

DETAILED DESCRIPTION:
This study is designed to test the association between cumulative fluids balance and ventilator associated events among critically ill patients.

Setting: This research will be carried out in four General Intensive Care Units at two hospitals in El Beheira Governorate, Egypt.

* For three months, from October 1, 2022 to January, 2023, all newly admitted mechanically ventilated patients who will fulfill the inclusion criteria and agree to participate will be screened on a daily basis.
* The investigators will calculate cumulative fluid balance as daily fluid balance within four days of the event of interest. Cumulative fluid balance will be computed as the sum of daily fluid balances over the previous 24 hours, calculated by total fluid input minus total fluid output on a specific day of ICU admission over the first four calendar days of mechanical ventilation. Insensible fluid loss, such as perspiration or evaporative water loss related to respiration will not be routinely assessed and will not be included in the calculation of cumulative fluid balance. The cumulative fluid balance from day 0 to day 1 will be labelled as day 1, and the following days as day 2 and day 3. Cumulative fluid balance at day 3 refers to the cumulative fluid balance during the first four calendar days.
* Variables associated with VAEs will be assessed for each patient including: age, gender, admission diagnosis, comorbidities; and ICU length of stay, APACH II score, Sofa score and duration of tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years,
* mechanically ventilated for ≥48 h and remain in the intensive care ≥4 days.

Exclusion Criteria:

* Patients with acute renal failure and needs dialysis,
* increasing daily minimum positive end-expiratory pressure (PEEP) or Fio2 during MV treatment
* hemodynamic instability

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: critically ill patients
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Ventilator-Associated Event | 7 days of mechanical ventilation
  VAEs classified as ventilator-associated complication (VAC), infection-related ventilator-associated complication (IVAC), or the possible ventilator-associated pneumonia (PVAP).

SECONDARY OUTCOMES:
Duration of MV | 7days
  Duration of mechanical ventilation
ICU length of stay | participants will be followed for the ICU length of stay, an expected average of 4 weeks
  ICU length of stay
ICU mortality | 28 day
  ICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Y Othman, Ass. Prof., Study Chair — Faculty of Nursing, Damanhour University
Locations (1):
- Faculty of nursing, Damanhūr, Behira, Egypt

REFERENCES:
- [Background] Unki P, Save S. Analysis of Fluid Balance as Predictor of Length of Assisted Mechanical Ventilation in Children Admitted to Pediatric Intensive Care Unit (PICU). Int J Pediatr. 2022 Mar 20;2022:2090323. doi: 10.1155/2022/2090323. eCollection 2022. PMID 35356099
- [Background] Wang W, Zhu S, He Q, Wang M, Kang Y, Zhang R, Ji P, Zou K, Klompas M, Zong Z, Sun X. Fluid Balance and Ventilator-Associated Events Among Patients Admitted to ICUs in China: A Nested Case-Control Study. Crit Care Med. 2022 Feb 1;50(2):307-316. doi: 10.1097/CCM.0000000000005227. PMID 34473657
- [Background] Chao WC, Chang WL, Wu CL, Chan MC. Using Objective Fluid Balance Data to Identify Pulmonary Edema in Subjects With Ventilator-Associated Events. Respir Care. 2018 Nov;63(11):1413-1420. doi: 10.4187/respcare.06221. Epub 2018 Aug 7. PMID 30087192
- [Background] Fang WF, Fang YT, Huang CH, Chen YM, Chang YC, Lin CY, Hung KY, Chang YT, Chen HC, Huang KT, Chang HC, Chen YC, Wang YH, Wang CC, Lin MC. Risk factors and associated outcomes of ventilator-associated events developed in 28 days among sepsis patients admitted to intensive care unit. Sci Rep. 2020 Jul 29;10(1):12702. doi: 10.1038/s41598-020-69731-3. PMID 32728165
- [Background] Klompas M, Branson R, Cawcutt K, Crist M, Eichenwald EC, Greene LR, Lee G, Maragakis LL, Powell K, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia, ventilator-associated events, and nonventilator hospital-acquired pneumonia in acute-care hospitals: 2022 Update. Infect Control Hosp Epidemiol. 2022 Jun;43(6):687-713. doi: 10.1017/ice.2022.88. Epub 2022 May 20. PMID 35589091